CLINICAL TRIAL: NCT04927494
Title: Promoting Cervical Cancer Screening Among African American and Sub Saharan African Immigrants
Brief Title: Cervical Cancer Prevention for Black Adults
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Adebola Adegboyega (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor-Investigator, Adebola Adegboyega, Assistant Professor, University of Kentucky
Organization: University of Kentucky (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Screening
Other Study IDs: 60704; K01CA251487 (NIH)
Record Dates: First submitted 2021-06-08; First posted 2021-06-16 (Actual); Last update posted 2025-06-29 (Actual); Status verified 2025-06

CONDITIONS: Cervical Cancer
Keywords: Cervical cancer screening; HPV self-sampling; African American; Sub-Saharan African immigrants
MeSH Terms: conditions — Uterine Cervical Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Black women cervical cancer screening (Experimental): Participants in this group with receive the Health is Wealth intervention.
  Interventions: Behavioral: Health is Wealth: A Cervical Health Program

INTERVENTIONS:
Behavioral: Health is Wealth: A Cervical Health Program — Health is Wealth: A Cervical Health Program will be introduced in a one-time 2-hour educational session, participants will be given HPV self-sampling kits, and instructional sheet that visually depicts the steps for self-sampling. The program will be culturally tailored to increase self-efficacy and knowledge while simultaneously addressing perceived health beliefs associated with cervical cancer and barriers associated with cervical cancer screening and HPV self-sampling. Content will be delivered in a group format (about 10-15 participants) by lecture, demonstration, and interactive exercises.

SUMMARY:
The goal of this study is to develop and pilot test an intervention, entitled Health is Wealth: A Cervical Health Program, designed to promote screening and reduce perceived barriers to Cervical Cancer (CC) screening.

Aim 1: Examine general awareness and cultural factors (fatalism, religiosity/spirituality, temporal orientation, medical mistrust, and acculturation) related to cancer control and prevention among African Americans (AA) and Sub Saharan African (SAI) Immigrants.

Aim 2: Examine the socioecological barriers and facilitators to CC screening and self-sampling to inform tailoring of an evidenced based cervical health program to promote CC screening.

Aim 3: Assess feasibility, acceptability, and preliminary efficacy in a pilot test of the Health is Wealth: A Cervical Health Program among 30 AA and 30 SAI women using quasi-experimental design.

This study will take place in 2 phases.

DETAILED DESCRIPTION:
In phase 1, the investigators will conduct a cross-sectional survey with 150 Black men and women to examine factors impacting cervical cancer screening. Also, as part of phase 1, Aim 2 employs focus groups and a quantitative Health Belief Model checklist with 30 participants to guide development of a tailored intervention. In phase 2, Aim 3 will assess feasibility, acceptability, and preliminary efficacy of the Health is Wealth: A Cervical Health Program intervention among 30 African American and 30 Sub-Saharan African immigrant women.

ELIGIBILITY:
Inclusion Criteria:

* Self-identify as Black woman (African American or Sub-Saharan African Immigrant)
* No pap smear within the last three years or no pap smear/HPV co-test within past five years
* Able to speak and write in English
* Reside in Kentucky

Exclusion Criteria:

* Do not self-identify as Black woman (African American or Sub-Saharan African Immigrant)
* History of hysterectomy
* History of cervical cancer
* Being pregnant
* Unable to speak and write in English
* Do not reside in Kentucky

Ages: 30 Years to 65 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Gender Based: Yes — Anatomically female with a cervix.
Enrollment: 60 (Actual)
Dates: Start 2023-01-01 (Actual); Primary Completion 2025-05-10 (Actual); Study Completion 2025-06-20 (Actual)

PRIMARY OUTCOMES:
Completion of HPV self-sampling | Baseline
  HPV self-sampling kit return
Change in Cervical cancer Knowledge | 6 months (Baseline, immediately post-test, 6 month follow up)
  Cervical cancer awareness will be assessed with Likert style questions (strongly disagree-1 to strongly agree-5) from the cervical cancer awareness toolkit. Awareness of warning signs and risk factors will be assessed with a prompted checklist. This instrument has been found to be valid and reliable in multiple populations.
Change in HPV knowledge | 6 months (Baseline, immediately post-test, 6 month follow up)
  Participants will complete 16 items assessing knowledge of HPV, 6 items about HPV testing, and 7 items about the vaccination. Response options included "True," "False," and "Don't know," with scoring allocating one point for each correct response, and zero points for incorrect or "Don't know" responses, summed across items, for a potential range of 0-29. This instrument has been found to be valid and reliable in multiple populations.
Change in Self-efficacy | 6 months (Baseline, immediately post-test, 6 month follow up)
  Self-efficacy will be assessed with 10 items measured on a five-point Likert-like scale response choices: strongly disagree (scores 1 point), disagree (scores 2point), neutral (scores 3 point), agree (scores 4 point) and strongly agree (scores 5 points), with higher scores indicating stronger feelings toward the construct. This is a well validated and reliable instrument.
Change in perceived barriers to screening | 6 months (Baseline, immediately post-test, 6 month follow up)
  Barriers will be assessed with 14 items measured on a five-point Likert-like scale response choices: strongly disagree (scores 1 point), disagree (scores 2point), neutral (scores 3 point), agree (scores 4 point) and strongly agree (scores 5 points), with higher scores indicating stronger feelings toward the construct

SECONDARY OUTCOMES:
Change in benefits | 6 months (Baseline, immediately post-test, 6 month follow up)
  Benefits will be assessed with 4 items measured on a five-point Likert-like scale response choices: strongly disagree (scores 1 point), disagree (scores 2 point), neutral (scores 3 point), agree (scores 4 point) and strongly agree (scores 5 points), with higher scores indicating stronger feelings toward the construct
Change in susceptibility | 6 months (Baseline, immediately post-test, 6 month follow up)
  Susceptibility will be assessed with 4 items measured on a five-point Likert-like scale response choices: strongly disagree (scores 1 point), disagree (scores 2 point), neutral (scores 3 point), agree (scores 4 point) and strongly agree (scores 5 points), with higher scores indicating stronger feelings toward the construct
Change in seriousness | 6 months (Baseline, immediately post-test, 6 month follow up)
  Seriousness will be assessed with 7 items measured on a five-point Likert-like scale response choices: strongly disagree (scores 1 point), disagree (scores 2 point), neutral (scores 3 point), agree (scores 4 point) and strongly agree (scores 5 points), with higher scores indicating stronger feelings toward the construct.

CONTACTS AND LOCATIONS:
Overall Officials: Adebola Adegboyega, PhD, Principal Investigator — University of Kentucky
Locations (1):
- University of Kentucky, Lexington, Kentucky, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Adegboyega A, Wiggins AT, Obielodan O, Dignan M, Schoenberg N. Beliefs associated with cancer screening behaviors among African Americans and Sub-Saharan African immigrant adults: a cross-sectional study. BMC Public Health. 2022 Nov 29;22(1):2219. doi: 10.1186/s12889-022-14591-x. PMID 36447190

DOCUMENTS (1):
  • Informed Consent Form (2024-10-15): https://cdn.clinicaltrials.gov/large-docs/94/NCT04927494/ICF_000.pdf